CLINICAL TRIAL: NCT07127861
Title: Effects of Treadmill-Based Gait Training in Patients With Stroke
Acronym: TreadmillACV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Salamanca (Other)
Collaborators: Colegio Profesional Fisioterapeutas Castilla y León (Unknown); INSTITUTO DE INVESTIGACION BIOMEDICA DE SALAMANCA (IBSAL) (Unknown)
Responsible Party: Principal Investigator, Marta Gómez Mateos, Physical therapist, University of Salamanca
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: INV-2025-58
Record Dates: First submitted 2025-08-10; First posted 2025-08-17 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Gait; Thermography; Walking Speed, Mesh id D000072797; Endurance; Step Time and Length; Gait Analysis

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial in which an intervention group will undergo treadmill training and the control group will not receive any intervention.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Experimental: Intervention Group TREADMILL GAIT TRAINING Participants will undergo a 15-minute treadmill gait training session using a safety harness and under the continuous supervision of a physiotherapist to ensure patient safety.
  The study will be carried out for 12 weeks with a frequency of two weekly sessions. During them, the participants will receive treadmill training.
  All participants will walk at a speed exceeding 2.5 km/h. The speed will be individually adjusted to provide a challenging yet appropriate intensity based on each participant's capabilities.
  Interventions: Other: Treadmill gait training
- No Intervention: Control Group (No Intervention): NO intervention

INTERVENTIONS:
Other: Treadmill gait training — Participants will undergo a 15-minute treadmill gait training session using a safety harness and under the continuous supervision of a physiotherapist to ensure patient safety. The study will be carried out for 12 weeks with a frequency of two weekly sessions. During them, the participants will receive treadmill training. All participants will walk at a speed exceeding 2.5 km/h. The speed will be individually adjusted to provide a challenging yet appropriate intensity based on each participant's capabilities.
  Arms: Intervention Group

SUMMARY:
Hemiplegia is one of the most common sequelae after stroke. Most patients develop thermal asymmetry between the affected and contralateral sides of the body, as well as an asymmetric gait pattern characterized by differences in the duration of gait cycle phases, step length, cadence, and weight distribution between limbs. These patterns result in reduced aerobic capacity, endurance, energy efficiency, and walking speed, negatively impacting the patient's functional abilities.

There are different methodologies for the treatment gait impairments. Among them, treadmill training has been investigated as an effective therapeutic approach to post-stroke rehabilitation.

Treadmill gait training may reduce asymmetry between hemibodies in hemiplegic patients.

For this reason, our aim is to describe the effects of treadmill training on gait, focusing on its impact on thermal asymmetry, walking speed, aerobic endurance, and the biomechanical and kinematic characteristics of gait.

Patients with hemiplegia will undergo treadmill-based gait training to evaluate its influence on the recovery of this sequel of stroke.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 80 years
* History of stroke at least six months prior
* Presence of hemiplegia or hemiparesis
* Ability to walk independently or with assistive devices

Exclusion Criteria:

* Cognitive impairments interfering with the understanding of treatment procedures
* Inability to get on and maintain position on the treadmill
* Severe heart failure
* Active inflammatory or infectious conditions at the time of evaluation
* Attendance below 80% of scheduled sessions

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-09-14 (Actual); Primary Completion 2025-09-15 (Actual); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Thermal asymmetry | 30 minutes
  Temperature and humidity will be recorded. Participants will arrive 15 minutes early for acclimatization, seated calmly in the assessment room, wearing shorts and without shoes or socks. They must avoid hot baths, creams, talcum powder, cosmetics, physical exercise, stimulants (caffeine, alcohol, nasal decongestants), smoking, and food intake (water allowed) within two hours prior. During this period, informed consent will be obtained and adhesive markers will be placed 1 cm laterally to the regions of interest: anterior thigh (5 cm above patella), anterior leg (5 cm below patella), posterosuperior leg (popliteal fossa), and posteroinferior leg (10 cm above heel).
  Thermal images will be taken in standing position (anterior and posterior views) and supine position (plantar surface), using a tripod-mounted camera at standardized distances and heights. For standing images, the camera will be positioned on a tripod at a distance of 2 m from the subject, at a height of 1

SECONDARY OUTCOMES:
Walking speed | 5 minutes
  The 10-Meter Walk Test (10MWT) will be used to evaluate walking speed. The test will be conducted in a hallway measuring more than 14 meters in length, with at least two meters available before the start line for acceleration and more than two meters after the finish line for deceleration.
Endurance | 30 minutes
  The 6-Minute Walk Test (6MWT) will be used to measure aerobic endurance. It is a submaximal cardiorespiratory effort test that measures the maximum distance a person can walk on a flat surface in six minutes. Before starting, the patient is instructed to walk as far as possible within six minutes, with the option to rest if needed. The evaluator starts the timer when the patient begins walking, pausing it during any rests and resuming when walking continues. Heart rate and oxygen saturation are recorded every minute, along with any pauses.
Gait Biomechanics and Kinematics | 10 minutes
  Gait biomechanics and kinematics will be measured through video recordings and analyzed using Kinovea software. Videos will be captured simultaneously from the frontal and sagittal planes while the patient walks along a marked corridor. Cameras mounted on tripods at a height of 70 cm will be positioned at designated points. The patient will walk back and forth between markers spaced one meter apart, ensuring they pass centrally between the markers in the frontal plane. Recordings will be made in slow motion to accurately observe lower limb movements for detailed biomechanical and kinematic analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Salamanca, Salamanca, Salamanca, Spain

IPD SHARING:
Plan to Share IPD: Yes
The study protocol and the CSR will be available from the publication of the results for 10 years in the repository of the University of Salamanca GREDOS.
Supporting Information: Study Protocol, CSR
Time Frame: From the publication of the results for 10 years
URL: http://gredos.usal.es/